CLINICAL TRIAL: NCT04599803
Title: Baseline Sleep Apnea Study #2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 102033
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea of Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Arm 1 (Experimental): Participants told they may have Obstructive Sleep Apnea (OSA) and provided a home sleep test (HST)
  Interventions: Device: Verily Sleep Apnea (VSA) Program/App

INTERVENTIONS:
Device: Verily Sleep Apnea (VSA) Program/App — The VSA program/app, is an Obstructive Sleep Apnea (OSA) management platform.

SUMMARY:
This is a single group, unblinded, prospective clinical study. This study seeks to understand patient diagnostic and treatment journey and positive airway pressure (PAP) therapy compliance for Verily Sleep Apnea (VSA) program/app users. Participants will enroll remotely and may undergo a home sleep test (HST). Upon confirmation of obstructive sleep apnea (OSA) and prescription of PAP therapy, the participant will begin using the VSA app to supplement PAP treatment. After 90 days of active participation, the participant will be given instructions for follow-up care, as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 or older
* Able to speak and read English
* Legal United States Resident with a Government Issued ID
* Participating in the Project Baseline Community Study
* Demonstrates understanding of the study requirements and is able and willing to sign the informed consent form
* Own a smartphone with a data plan and be the primary user of the smartphone; smartphone must use Android Lollipop (5.1+/ API 22+) or iOS 11.X+
* Own a computer with a web camera
* Consistent access to electricity and wifi for the duration of the study
* Have a high risk of OSA as determined by screening questionnaire
* Good candidate for PAP therapy, in the opinion of the managing clinician
* Without significant limitation in ability to participate in the study, in the opinion of the investigator.

Exclusion Criteria:

* Previously diagnosed with sleep apnea or other sleep disorders, that in the opinion of the investigator, makes the participant ineligible (e.g., Obstructive Sleep Apnea, Central Sleep Apnea, Complex Sleep Apnea, chronic insomnia)
* Participant is a shift worker (indicated by having a night shift schedule on a regular basis, or a work shift that changes or rotates on a daily, weekly, or monthly basis)
* Sponsor employees and individuals working on Project Baseline
* Self reported to be pregnant or planning to become pregnant during the study period
* Current use of home oxygenation devices, such as supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Sullivan, MD, Principal Investigator — Verily Life Sciences LLC
Locations (1):
- Verily Life Sciences LLC, South San Francisco, California, United States

REFERENCES:
- [Derived] Kumar S, Rudie E, Dorsey C, Caswell K, Blase A, Sert Kuniyoshi F, Benjafield AV, Sullivan SS. Pilot study of positive airway pressure usage, patient journey and program engagement for users of a digital obstructive sleep apnea program. Front Digit Health. 2023 Jun 7;5:1043578. doi: 10.3389/fdgth.2023.1043578. eCollection 2023. PMID 37351372
- [Derived] Kumar S, Rudie E, Dorsey C, Blase A, Benjafield AV, Sullivan SS. Assessment of Patient Journey Metrics for Users of a Digital Obstructive Sleep Apnea Program: Single-Arm Feasibility Pilot Study. JMIR Form Res. 2022 Jan 12;6(1):e31698. doi: 10.2196/31698. PMID 34792470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted entirely virtually using the Baseline Platform, a comprehensive remote clinical studies platform for recruitment, consenting, screening, enrollment, data collection, and study monitoring.
Pre-assignment Details: Participants must have met all eligibility criteria and logged into the Verily Sleep Apnea (VSA) App in order to be considered enrolled.
Period: Overall Study
Arm/Group | Arm 1
Started | 187 (Defined for the purpose of this table to have met eligibility criteria and signed into the Verily Sleep Apnea (VSA) app)
Completed | 156
Not Completed | 31
Not completed — Withdrawal by Subject | 5
Not completed — Lost to Follow-up | 26

BASELINE CHARACTERISTICS:
Population: Participants that were diagnosed with sleep apnea and prescribed a positive airway pressure (PAP) device
Groups:
- Participants Diagnosed With Obstructive Sleep Apnea: This will be a single arm study of participants that are diagnosed with Obstructive Sleep Apnea (OSA) during the study. Upon confirmation of OSA and prescription of positive airway pressure (PAP) therapy, the participant will begin using the Verily Sleep Apnea (VSA) app to supplement PAP treatment.
  Verily Sleep Apnea (VSA) Program/App: The VSA program/app, is an Obstructive Sleep Apnea (OSA) management platform.
Arm/Group | Participants Diagnosed With Obstructive Sleep Apnea
Number analyzed (Participants) | 105
Age, Categorical [Count of Participants; unit: Participants] — Population: Only participants that were prescribed a PAP device were included evaluable population for analysis.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 96
    >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Only participants that were prescribed a PAP device were included evaluable population for analysis.
  Years | 48 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only participants that were prescribed a PAP device were included evaluable population for analysis.
  Participants
    Female | 61
    Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only participants that were prescribed a PAP device were included evaluable population for analysis.
  Participants
    Hispanic or Latino | 25
    Not Hispanic or Latino | 0
    Unknown or Not Reported | 80
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Only participants that were prescribed a PAP device were included evaluable population for analysis.
  Participants could select all that apply, so percentages sum to more than 100%.
  Participants
    American Indian or Alaska Native | 1
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 73
    More than one race | 27
    Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: Only participants that were prescribed a PAP device were included evaluable population for analysis.
  Participants
    United States | 105

OUTCOME MEASURES:

1. Primary Outcome: Time (Number of Days) From When Participant is Told They May Have OSA to When They Receive HST Prescription
Description: Time (number of days) from when participant is told they may have OSA to when they receive HST prescription
Time Frame: 147 Days
Population: Participants told they may have Obstructive Sleep Apnea (OSA) and provided a home sleep test (HST)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1
Number analyzed (Participants) | 157
days | 7.4 (2.7)

2. Primary Outcome: Time (Number of Days) From When Participant Receives HST Prescription to When They Receive Their Diagnosis
Description: Time from when the participant receives HST prescription to OSA diagnosis.
Time Frame: 164 days
Population: Participants diagnosed with OSA
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1
Number analyzed (Participants) | 114
days | 13.9 (9.6)

3. Primary Outcome: Time (Number of Days) From OSA Diagnosis to PAP Therapy Initiation
Description: Time from OSA diagnosis to PAP therapy initiation.
Time Frame: 153 Days
Population: Participants diagnosed with OSA and received PAP device
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1
Number analyzed (Participants) | 105
days | 8.1 (9.3)

4. Primary Outcome: Time (Number of Days) From Therapy Initiation to When 90-day Compliance Threshold is Achieved
Description: Time (number of days) from therapy initiation to when 90-day compliance threshold is achieved.
  90-day Compliance is defined as ≥ 4 hours per night on 70% of nights during a consecutive 30 day period anytime during the first 90 days.
Time Frame: 90 Days
Population: Participants who reached compliance with their PAP device
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm 1
Number analyzed (Participants) | 68
days | 37.5 (14.25)

5. Secondary Outcome: Completion Rates Among Individuals Who Had an HST Ordered
Description: Among individuals prescribed a HST, % of individuals who completed the HST and had interpretable results.
Time Frame: 161 Days
Population: Participants who received a HST
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 157
Participants | 153

6. Secondary Outcome: Completion Rates Among Individuals Prescribed a PAP Device
Description: Among individuals prescribed a PAP device, % of individuals who filled the order (PAP device delivered to them).
Time Frame: 153 Days
Population: Participants diagnosed with OSA who received a prescription for PAP as part of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 105
Participants | 105

7. Secondary Outcome: Completion Rates Among Individuals Prescribed a PAP Device
Description: Percentage of individuals who used the PAP device at least once during the 90 days
Time Frame: 90 Days
Population: Participants diagnosed with OSA and received PAP device
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 105
Participants | 103

8. Secondary Outcome: Percent of Participants Who Meet 90 Day Compliance Success Criteria
Description: Compliance Metrics - Percent of participants who meet 90 day compliance success criteria, as defined by: ≥ 4 hours per night on 70% of nights during a consecutive 30 day period anytime during the first 90 days
Time Frame: 90 Days
Population: Participants diagnosed with OSA and received PAP device
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1
Number analyzed (Participants) | 105
Participants | 68

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire duration of participation (232 Days). Reported Adverse Events were monitored through study completion.
Description: Per Protocol:
  An Adverse Event (AE) is defined as any untoward medical occurrence, unintended disease or injury in subjects, users or other persons, that is considered a change from baseline or pre-study status, whether or not related to the investigational medical device.
Groups:
- Arm 1: Participants diagnosed with Obstructive Sleep Apnea (OSA) and provided a positive airway pressure (PAP) device.
  This was a single arm study of participants that are diagnosed with Obstructive Sleep Apnea (OSA) during the study. Upon confirmation of OSA and prescription of positive airway pressure (PAP) therapy, the participant began using the Verily Sleep Apnea (VSA) app to supplement PAP treatment.
Arm/Group | Arm 1
All-Cause Mortality (participants affected / at risk) | 0/105
Serious Adverse Events (participants affected / at risk) | 1/105
Other Adverse Events (participants affected / at risk) | 14/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=105)
Hospitalization subsequent to apparent syncopal event leading to chest wall injury (Injury, poisoning and procedural complications) | 1 (1) — Hospitalization subsequent to apparent syncopal event leading to chest wall injury
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=105)
Skin Sore (Skin and subcutaneous tissue disorders) | 1 (1)
Tooth Pain (Injury, poisoning and procedural complications) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Fatigue and sore throat due to COVID-19 (Infections and infestations) | 1 (1)
Sinus Infection (Infections and infestations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Kidney Stone Pain (Renal and urinary disorders) | 1 (1)
Cough due to COVID-19 (Infections and infestations) | 1 (1)
Respiratory illness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough and upper respiratory symptoms due to COVID-19 (Infections and infestations) | 1 (1)
Fever due to COVID-19 (Infections and infestations) | 1 (1)
Congestion due to COVID-19 (Infections and infestations) | 1 (1)
Nausea/ Diarrhea (General disorders) | 1 (1)
Dry nose/bloody nose due to weather (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT04599803/Prot_SAP_001.pdf